CLINICAL TRIAL: NCT01763957
Title: The Effectiveness of Circular Muscle Exercise (the Paula Method) as Compared to Pelvic Floor Muscle Training (PFMT), for Urinary Stress Incontinence (SUI) in Menopausal Women: A Randomized Controlled Trial
Brief Title: Paula Method Compared to Pelvic Floor Muscle Training (PFMT), for Urinary Stress Incontinence
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Paula/PFMT-HMO-CTIL
Record Dates: First submitted 2012-12-17; First posted 2013-01-09 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2012-12

CONDITIONS: Stress Urinary Incontinence; Sexual Satisfaction; Quality of Life
MeSH Terms: conditions — Urinary Incontinence, Stress; Orgasm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pelvic Floor Muscle Training (PFMT) (Active Comparator)
  Interventions: Behavioral: Pelvic Floor Muscle Training (PFMT)
- Paula Method (Active Comparator)
  Interventions: Behavioral: Paula Method

INTERVENTIONS:
Behavioral: Paula Method — All subjects allocated to this group will receive one group lesson, 45 minute sessions once a week for twelve weeks. All will be encouraged to practice daily for 15-45 minutes at home. The teachers will be followed a set exercise list.
  Arms: Paula Method
Behavioral: Pelvic Floor Muscle Training (PFMT) — All subjects allocated to this group will receive one group lesson, 45 minute sessions once a week for twelve weeks. All will be encouraged to practice daily for 15-45 minutes at home. The teachers will be followed a set exercise list .
  Arms: Pelvic Floor Muscle Training (PFMT)

SUMMARY:
The Investigators decided to examine whether the Paula method is more effective than Pelvic Floor Muscle Training (PFMT) in terms of urinary leakage amount, as it measured by pad test in menopause women without an hormonal therapy. In addition to the pad test and two urinary incontinence questionnaires, we will use other assessment tools such as; quality of life and sexual function which have been found to correlate significantly with pad test results. These results may indicate that menopausal women with Stress Urinary Incontinence may be more successful controlling incontinence if they will practice the Paula method as compared to PFMT.

ELIGIBILITY:
Inclusion Criteria:

* women after menopause (12 months with no period)
* aged 40 or more
* have a positive pad test leakage of 1-50 grams
* no systemic or local hormonal therapy
* literate in Hebrew and/or English

Exclusion Criteria:

* women suffering from illnesses which limit physical activity (cardiac, respiratory, psychiatric or neurological disorders)
* pelvic surgery within the last 6 months
* post hysterectomy or oophorectomy genital prolapse grade 3 or higher

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
change in the quantity of urinary leakage, measured by the one hour pad test | 1) Baseline 2) After 12 weeks of exercise intervention 3) 12 months after completion of the intervention
  To examine whether the Paula method intervention is more effective than PFMT in reducing urinary leakage in menopausal women with SUI

SECONDARY OUTCOMES:
change in the urinary leakage questionnaires, measured by ICIQ-UI and QUID | 1) Baseline 2) After 12 weeks of exercise intervention 3) 12 months after completion of the intervention
improvement of sexual function | 1) Baseline 2) After 12 weeks of exercise intervention 3) 12 months after completion of the intervention
  To evaluate the effectiveness of both methods to improve sexual function in women diagnosed with SUI
improvement of quality of life | 1) Baseline 2) After 12 weeks of exercise intervention 3) 12 months after completion of the intervention
  To evaluate the effectiveness of both methods to improve quality of life in women diagnosed with SUI

CONTACTS AND LOCATIONS:
Overall Officials: Drorith Hochner-Celnikier, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel